CLINICAL TRIAL: NCT06976736
Title: A Long-term Follow-up Study to Assess Safety in Participants Who Received an Investigational T-Cell Receptor Engineered T-Cell (TCR-T) Product
Brief Title: A Long Term Follow-up Study of TScan TCR-T Products
Acronym: LTFU
Status: Recruiting | Type: Observational
Sponsor: TScan Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TSCAN-004
Record Dates: First submitted 2025-04-18; First posted 2025-05-16 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: AML; ALL; MDS
Keywords: TSCAN; Cell Therapies; TCR-T Cell Therapy; Long Term Follow-Up (LTFU); TSC-101; TSC-100; TSCAN-001
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Approximately 20 ml of whole blood will be collected at each visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: No study drug will be administered during this trial. Participants previously treated with TSC-100 or TSC-101 in a TScan study will be evaluated for long-term safety and efficacy.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Long Term Follow-Up for participants treated with TSC-100 or TSC-101 TCR-T products

SUMMARY:
The purpose of this Long-Term Follow-Up (LTFU) study is to monitor participants who have previously received TSC-100 or TSC-101 TCR-T therapies in the TSCAN-001 study. Participants will be monitored for 15 years from the date of TCR-T cell therapy administration to assess long-term safety and efficacy.

DETAILED DESCRIPTION:
Participants will enroll in this LTFU study after completing the TSCAN-001 interventional trial. No additional study drug will be administered; however, participants may receive other cancer treatments as needed while being monitored for long-term safety.

Enrollment will occur after completion of the TSCAN-001 study, and participants will be monitored for safety and efficacy over a 15 year period.

ELIGIBILITY:
Inclusion Criteria:

* Participants who received a TCR-T cellular therapy in a clinical study sponsored by TScan Therapeutics.
* Signed informed consent.

Exclusion Criteria:

* None

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who received TSC-100 or TSC-101 cellular therapies.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-09-09 (Estimated); Primary Completion 2040-09 (Estimated); Study Completion 2040-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | 15 years post TCR-T administration
  To assess the long-term safety of TSC-100 and TSC-101 in participants by evaluating the incidence, duration, and outcome of adverse events and adverse events of special interest.

SECONDARY OUTCOMES:
Overall Survival | 15 years post TCR-T administration
  To asses the long-term efficacy of TSC-100 and TSC-101 in participants by evaluating:
  Overall survival (OS) is defined as the time interval between the date of stem cell transplant or TCR-T cell infusion and death for any cause.
Relapse-free survival | 15 years post TCR-T administration
  To asses the long-term efficacy of TSC-100 and TSC-101 in participants by evaluating:
  Relapse-free survival (RFS) is defined as the time from date of transplant in the parent study to death or relapse, whichever comes first.
Progression-free survival | 15 years post TCR-T administration
  To asses the long-term efficacy of TSC-100 and TSC-101 in participants by evaluating:
  Progression-free survival (PFS) is defined as the time from date of first TCR-T cell infusion in the parent study to death or disease progression, whichever comes first.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Matzko, MD, Study Director — Medical Monitor
Locations (2):
- United States (2):
  - City of Hope, Duarte, California
  - Mount Sinai, New York, New York

IPD SHARING:
Plan to Share IPD: No